CLINICAL TRIAL: NCT05390593
Title: Treatment for Major Depressive Disorder With Intermittent Theta-burst Stimulation: a Three-track Approach in Affective Computing, Randomized Controlled Trial, and Meta-analysis
Brief Title: Treatment for Major Depressive Disorder With Intermittent Theta-burst Stimulation
Acronym: iTBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chih-Wei Hsu, Psychiatry Department, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMRPG8L0871
Record Dates: First submitted 2022-04-13; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Repetitive transcranial magnetic stimulation; Mood Disorders
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- iTBS-1800 (Experimental): The active group will receive 1800 pluse of intermittent theta-bursts in the left dorsolateral prefrontal cortex.
  Interventions: Device: iTBS-1800
- iTBS-1200 (Experimental): The active group will receive 1200 pluse of intermittent theta-bursts in the left dorsolateral prefrontal cortex.
  Interventions: Device: iTBS-1200

INTERVENTIONS:
Device: iTBS-1800 — Participants in the 1800-pulse intermittent TBS (iTBS-1800) active stimulation group will receive three-pulse 50-Hz pulses for 2 weeks at an intensity of 80% active motor threshold (MT) to Left DLPFC, twice a day. Stimulation will use a MAG & More stimulator.
  Arms: iTBS-1800
Device: iTBS-1200 — Participants in the 1200-pulse intermittent TBS (iTBS-1200) active stimulation group will receive three-pulse 50-Hz pulses for 2 weeks at an intensity of 80% active motor threshold (MT) to Left DLPFC, twice a day. Stimulation will use a MAG & More stimulator.
  Arms: iTBS-1200

SUMMARY:
The main purpose of this study is to investigate the two different intermittent Theta Burst (iTBS) repetitive transcranial magnetic stimulation (rTMS), its effectiveness in alleviating depressive symptoms. All patients are randomized to two different iTBS groups.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of major depressive disorder according to DSM-5
2. Total HAM-D17 score of greater than or equal to 18 and Item 3 score less than 4 at screening visit. CGI-S score less than 4.
3. Before treatment, patient have to stop antidepressant for at least 1 weeks.
4. Capable and willing to provide informed consent.

Exclusion Criteria:

1. Have a concomitant major, unstable medical or neurologic illness :

   * Psychiatric disorder: Schizoprenia, Bipolar disorder, Obsessive Compulsive Disorder, Posttraumatic Stress Disorder, substance use disorder.
   * Severe brian disease: Brain tumor, encephalitis, brian injury.
2. Intracranial implant and other ferromagnetic materials close to the head.
3. History of Seizures.
4. Cardiac pacemaker.
5. Pregnancy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in 17-item Hamilton Depression Rating Scale | Baseline, Week 1, Week 2, Week 4
  17-item Hamilton Depression Rating Scale (range from 0 to 52 with higher scores indicating more depression)
Change in Montgomery-Asberg Depression Rating Scale | Baseline, Week 1, Week 2, Week 4
  Montgomery-Asberg Depression Rating Scale (range from 0 to 54 with higher scores indicating more depression)
Change in Beck Anxiety Inventory | Baseline, Week 1, Week 2, Week 4
  Beck Anxiety Inventory (range from 0 to 63 with higher scores indicating more severe anxitey)

SECONDARY OUTCOMES:
Response rate after 2-week treatment at the end of iTBS (HDRD-17 ) | Baseline, Week 1, Week 2, Week 4
  Improvement > 50 % of HDRD-17
Response rate after 2-week treatment at the end of iTBS (MADRS) | Baseline, Week 1, Week 2, Week 4
  Improvement > 50 % of MADRS
Changes in Clinical Global Index Severity | Baseline, Week 1, Week 2, Week 4
  Clinical Global Index
Changes in Heart Rate Variability (HRV) band | Baseline, Week 1, Day 3, Week 2, Week 4
  Heart rate variability measured by Wegene 8Z11
Changes in EEG band | Baseline, Week 1, Day 3, Week 2, Week 4
  Changes in EEG band before and after brain stimulation. Subject EEG activity including EEG waveform, spectrum, spectrogram, and power in the slow (0.1-1 Hz), delta (1 to 4 Hz), theta (4 to 8 Hz), alpha (8 to 12 Hz), beta (12 to 25 Hz), and gamma (25 to 70 Hz) bands.
Change in BDNF | Baseline, Week 2
  Changes in BDNF values
Change in TSH | Baseline, Week 2
  Change in TSH values
Change in T3 | Baseline, Week 2
  Change in T3
Change in T4 | Baseline, Week 2
  Change in T4
Change in cortisol | Baseline, Week 2
  Change in cortisol

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGungMH, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No